CLINICAL TRIAL: NCT06881602
Title: Remote Clinical Monitoring After Robotic Distal Pancreatectomy: a Pilot and Feasibility Study
Brief Title: Remote Clinical Monitoring After Robotic Distal Pancreatectomy
Acronym: TOTEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Professor, Dr, Jessa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/012
Record Dates: First submitted 2025-02-27; First posted 2025-03-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Digital Health
Keywords: Remote monitoring; Pancreatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote clinical monitoring (Experimental): The application of remote clinical monitoring after a distal robotic pancreatectomy
  Interventions: Procedure: Remote clinical monitoring

INTERVENTIONS:
Procedure: Remote clinical monitoring — Patients after a distal pancreatectomy will be discharged faster from the hospital and will be remote monitored

SUMMARY:
This feasibility trial has three main objectives:

* To investigate the impact of the transmural care pathway TOTeM on the Length of Stay (LOS) for patients undergoing robotic distal pancreatectomy.
* To investigate the feasibility of the implementation of TOTeM for patients undergoing robotic distal pancreatic surgery, we will measure the recruitment rate by tracking the number of eligible patients who are approached for participation, the percentage who consent to join the study over a specified time period, and the adherence rate which describes how well participants follow the study protocol including the prescribed interventions or follow-up assessments.
* Assessment of the potential changes in medical costs and outcomes for the purpose of performing a cost-effectiveness analysis from a hospital and patient perspective.

DETAILED DESCRIPTION:
Due to fast progress and improvements in robotic surgery, minimally invasive procedures for complex surgery have become increasingly feasible for the vast majority of patients. Over recent years, minimally distal pancreatectomy (MDP) has become the preferred approach for distal pancreatectomy. This minimally invasive alternative offers less postoperative pain, better cosmetic outcomes, a quicker recovery, a shorter hospital stay, decreased morbidity, reduced intraoperative blood loss, and reduced health care costs. This shift in care models has enabled patients to return home more quickly after surgery, while their recovery continues to be closely monitored.

Hospitals are increasingly confronted with high bed occupancy rates and the need to use staff more efficiently. This has emphasized the importance of optimizing the length of stay for patients undergoing pancreatectomy, ensuring they can be discharged sooner without compromising their recovery. Early discharge from the hospital, combined with remote monitoring, offers a promising solution to these challenges. Thanks to advances in technology, patients can be monitored remotely after discharge by healthcare professionals allowing for early detection of potential complications and timely intervention, all while the patient recovers in the comfort of their own home. This approach also facilitates the effective implementation of transmurally coordinated care pathways (care delivered across different levels of the healthcare system), ensuring seamless communication and care transitions between hospital and home.

The TOTeM (Transmurale Opvolging met TeleMonitoring na chirurgie) project, supported by the Federale Overheidsdienst Volksgezondheid, Veiligheid van de Voedselketen en Leefmilieu, focuses on remote monitoring of patients with the help of wearable monitoring devices and a telemonitoring hub. Unlike the current approach where the patient is admitted to the intensive care unit (ICU) after surgery, patients will be immediately transferred to the ward. The patient is sent home after surgery as early as medically possible (as defined by reaching all of the time to be fit criteria), with qualitative and specialized follow-up in the home setting. The time to be fit criteria include: oral pain medication only, independent walking, oral intake, hemodynamically (90% of baseline blood pressure, heart rate in 90% of normal range) and respiratory (no need for extra oxygen) stable, and no drains or urinary catheters. After discharge, the patient is contacted by the telemonitoring hub through a daily videocall. Parameters are assessed up to three times a day. Follow-up via the mobile application and videocall is foreseen up to ten days postoperatively. The telemonitoring hub screens all input from the questionnaires completed by the patient as well as the parameters that are obtained via wearable monitoring devices. If necessary, the patient is contacted or an escalation protocol is triggered. The project aims to enable a faster recovery of patients in a familiar home environment and a more active role of the patient in their recovery process. For the hospital, the faster discharge offers the opportunity to optimize bed occupancy. On a societal level, the social cost of care may decrease.

This pilot and feasibility study focuses on the application of remote clinical monitoring following robotic distal pancreatectomy. By evaluating the feasibility and effect of the implementation of such a care model, this research aims to contribute to optimizing care for patients undergoing these complex procedures, while also alleviating pressure on hospital resources and staff.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Competent to provide informed consent
* Fluent in Dutch
* Cognitively capable of understanding and engaging with the study
* Undergoing robotic distal pancreatectomy
* Owing a smartphone or has a caregiver who can assist
* Does not live alone
* Have a valid national identification number

Exclusion Criteria:

* Extended left pancreatectomy
* Spleen-preserving procedure
* Residing in a nursing home
* Patients who are deemed unsuitable for the study by the physician based on clinical evaluation
* Absence of informed consent or request to not participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of stay in hospital | during hospital stay, an average of 4 days
  The primary outcome measurement for the TOTeM care pathway in patients undergoing robotic distal pancreatectomy is the length of stay, which is the total time measured from day of surgery to the day of hospital discharge

SECONDARY OUTCOMES:
Evaluation of the recruitment rate | during whole study period, an average of 1 year
  The feasibility of this pilot study is assessed by means of the recruitment rate, defined by the number of eligible patients who are approached for participation and the percentage who consent to join the study over a specified time period. The recruitment rate is defined as excellent if 20 patients can be enrolled in this study in one year.
Evaluation of the adherence rate | during whole study period, an average of 1 year
  The feasibility of this pilot study is assessed by the adherence rate, which describes how well participants follow the study protocol including the prescribed interventions or follow-up assessments. The adherence rate is defined as excellent if ≥80% of the patients followed the study protocol including the prescribed interventions or follow-up assessments.
Evaluation of medical costs | during study time of patient, an average of 3 months
  Evaluation of the potential changes in medical costs for the hospital and for the individual patient
Assessment of surgical fear | At baseline
  The short and long term surgical fear questionnaire will be evaluated at baseline, before the surgery. The short and long term questionnaire consist each of 4 questions, where 0 indicates no fear and 10 indicates extreme fear.
Quality of Life: EQ5D Questionnaire | at baseline (day of surgery), Day7, Day28, Month3
  Questionnaire measuring patients' general health and quality of life: EQ5D = EuroQol-5 Dimensions: mobility, self-care, daily activities, pain/discomfort, anxiety/depression. A score of 0 represent a very low quality of life, where score of 1 represents the maximum score.
Quality of Life: SF-36 Questionnaire | at baseline, Day 7, Day 28, Month 3
  This questionnaire contains 36 questions and 8 dimensions: physical functioning, physical limitations, mental functioning, emotional limitations, social functioning, pain, general health, vitality. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Evaluation of the technology acceptance questionnaire | baseline
  Evaluation of the technology acceptance questionnaire, which contains 17 statements where patient can (completely) disagree, no opion or (completely) agree with.
Pain scores (numerical rating scales) | 3 times per day for 10 days after the surgery
  Evaluation of different pain scores (abdominal pain, lower abdominal pain, pain at wound stitch hole, shoulder pain and pain after eating). These are numerical rating scales with 0 having no pain at all and 10 having extreme pain.
Satisfaction of patients | on day 10 after the surgery
  * Degree to which the patient is satisfied with the care pathway, felt safe during remote monitoring, and if they received sufficient information about the follow-up period.
  * Measured with Numeric Rating Scale (NRS), with 0 not satisfied at all and 10 extremely satisfied
Evaluation of pain medication | daily up to 10 days after surgery
  Assessment of the number of pain medication taken every day after the surgery
Evaluation of the acceptability of the remote care pathway | on postoperative day 10
  This wil be evaluated with a validated questionnaire containing 8 statements which the patient need to score as (completely) agree, no opinion or (completely) disagree
Evaluation of study patients admitted to the ICU | during study period, an average of 1 year
  The number of patients admitted to the ICU after surgery will be assessed
Evaluation of unplanned medical consultations or visits | during study period of the patient, an average of 3 months
  Assessment of unplanned readmission rate and/or unscheduled home visits from a general practitioner or other medical doctor and/or emergency consultations
Evaluation of post-operative complicatons | during study period of the patient, an average of 3 months
  Assessment of post-operative complications associated with distal pancreatectomy
Evaluation of respiratory rate | during 10 days after surgery
  Assessment of the respiratory rate, defined in breaths per minute.
Evaluation of the Intervention Appropriateness Measure | on postoperative day 10
  This wil be evaluated with a validated questionnaire containing 8 statements which the patient need to score as (completely) agree, no opinion or (completely) disagree
Evaluation of the Feasibility of Intervention Measure | on postoperative day 10
  This wil be evaluated with a validated questionnaire containing 8 statements which the patient need to score as (completely) agree, no opinion or (completely) disagree
Evaluation of temperature | during 10 days after surgery
  Assessment of the temperature of the patient, defined in °C.
Evaluation of oxygen saturation in blood | during 10 days after surgery
  Assessment of oxygen saturation in blood, measured in %